CLINICAL TRIAL: NCT05931094
Title: Effects of Augmented Reality Game-based Training on Social Communication of Children With Autism Spectrum Disorder
Brief Title: Augmented Reality Game-based Training on Social Communication of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F723 - Project B
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Augmented Reality; Social communication
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR group (Experimental): Augmented Reality based games
  Interventions: Other: Augmented Reality based games
- Traditional therapy group (Active Comparator): Traditional therapy
  Interventions: Other: Traditional therapy

INTERVENTIONS:
Other: Augmented Reality based games — Games of Wonder Tree Augmented Reality
  Arms: AR group
Other: Traditional therapy — Traditional therapy based on play activities utilizing blocks, colors, Velcro-based toys.
  Arms: Traditional therapy group

SUMMARY:
The study aims to determine the effects augmented reality game-based training on social communication of children with autism spectrum disorder.

DETAILED DESCRIPTION:
Augmented Reality allows children to see a representation of imaginary content and pretend play overlaid on the real-world environment. Today, technology can be a safe and motivating way of engaging children with autism in social interaction activities. Current research in therapeutic technology for autism is aimed toward improving behavior and psychomotor activities that impact social communication. The aim of this research project is to help teachers, parents, practitioners, and researchers to understand the unique strengths of their children with autism along with technology based educational and therapeutic activities for home and classroom.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with autism spectrum disorder in the age range of 5-12 years at verbal imitation and 1-step command following.

Exclusion Criteria:

* Sensory issues and patients on medication.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale | After 8 weeks
  The Social Responsiveness Scale, Second Edition (SRS-2) measures social ability of children to adults. It is used primarily with individuals on the autism spectrum, family members of individuals on the autism spectrum, and others who have social impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Child Development Center, Islamabad, AL, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berenguer C, Baixauli I, Gomez S, Andres MEP, De Stasio S. Exploring the Impact of Augmented Reality in Children and Adolescents with Autism Spectrum Disorder: A Systematic Review. Int J Environ Res Public Health. 2020 Aug 24;17(17):6143. doi: 10.3390/ijerph17176143. PMID 32847074
- [Background] Liu R, Salisbury JP, Vahabzadeh A, Sahin NT. Feasibility of an Autism-Focused Augmented Reality Smartglasses System for Social Communication and Behavioral Coaching. Front Pediatr. 2017 Jun 26;5:145. doi: 10.3389/fped.2017.00145. eCollection 2017. PMID 28695116